CLINICAL TRIAL: NCT01055080
Title: Pilot Study of Dietary Prevention of Type 1 Diabetes Associated Beta-cell Autoimmunity in Children at Genetic Risk
Brief Title: Insulin-free Cow Milk Formula in Prevention of Type 1 Diabetes Associated Autoimmunity - FINDIA Pilot Study
Acronym: FINDIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Collaborators: Valio Ltd (Industry); University of Turku (Other); University of Helsinki (Other); University of Eastern Finland (Other)
Responsible Party: Outi Vaarala, National Institute for Health and Welfare, Finland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FINDIA2002
Record Dates: First submitted 2010-01-22; First posted 2010-01-25 (Estimated); Last update posted 2010-01-25 (Estimated); Status verified 2010-01

CONDITIONS: Beta-cell Autoimmunity
Keywords: type 1 diabetes; beta-cell autoantibodies; cow's milk formula; bovine insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cow's milk formula (Placebo Comparator)
  Interventions: Dietary Supplement: Cow's milk formula
- Bovine insulin-free whey based formula (Active Comparator)
  Interventions: Dietary Supplement: Cow's milk formula
- Whey-based hydrolysed formula (Active Comparator)
  Interventions: Dietary Supplement: Cow's milk formula

INTERVENTIONS:
Dietary Supplement: Cow's milk formula — Weaning to three different type of cow's milk formula when breast milk is not available during the first 6 months of life

SUMMARY:
The purpose of this study is to determine whether weaning to whey-based hydrolysed formula or essentially bovine insulin free whey-based FINDIA formula instead of standard cow's milk based formula is effective in the prevention of type 1 diabetes associated beta-cell autoimmunity in children at genetic risk of type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* HLA-conferred genetic susceptibility for type 1 diabetes

Exclusion Criteria:

* Pre-term, maternal diabetes with insulin treatment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 987 (Actual)
Dates: Start 2002-05; Primary Completion 2006-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Beta-cell autoantibodies | 3,6,12,24,36,48,60,72 months

CONTACTS AND LOCATIONS:
Overall Officials: Outi Vaarala, MD PhD, Principal Investigator — Finnish Institute for Health and Welfare

REFERENCES:
- [Derived] de Goffau MC, Luopajarvi K, Knip M, Ilonen J, Ruohtula T, Harkonen T, Orivuori L, Hakala S, Welling GW, Harmsen HJ, Vaarala O. Fecal microbiota composition differs between children with beta-cell autoimmunity and those without. Diabetes. 2013 Apr;62(4):1238-44. doi: 10.2337/db12-0526. Epub 2012 Dec 28. PMID 23274889
- [Derived] Vaarala O, Ilonen J, Ruohtula T, Pesola J, Virtanen SM, Harkonen T, Koski M, Kallioinen H, Tossavainen O, Poussa T, Jarvenpaa AL, Komulainen J, Lounamaa R, Akerblom HK, Knip M. Removal of Bovine Insulin From Cow's Milk Formula and Early Initiation of Beta-Cell Autoimmunity in the FINDIA Pilot Study. Arch Pediatr Adolesc Med. 2012 Jul 1;166(7):608-14. doi: 10.1001/archpediatrics.2011.1559. PMID 22393174